CLINICAL TRIAL: NCT04241185
Title: A Phase 3, Randomized, Double-blind, Placebo-controlled Clinical Trial to Study the Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Chemoradiotherapy (CRT) Versus CRT Alone in Participants With Muscle-invasive Bladder Cancer (MIBC) (KEYNOTE-992)
Brief Title: Efficacy and Safety of Pembrolizumab (MK-3475) in Combination With Chemoradiotherapy (CRT) Versus CRT Alone in Muscle-invasive Bladder Cancer (MIBC) (MK-3475-992/KEYNOTE-992)
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 3475-992; MK-3475-992 (Other: MSD); 205383 (Registry Identifier: JAPIC-CTI); U1111-1287-4190 (Other: UTN); 2023-503500-87 (Registry Identifier: EU CT); jRCT2080225287 (Registry Identifier: jRCT); 2019-004023-20 (EudraCT Number)
Record Dates: First submitted 2020-01-22; First posted 2020-01-27 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-11

CONDITIONS: Urinary Bladder Neoplasms
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — pembrolizumab; Cisplatin; Fluorouracil; Mitomycin; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: All Sponsor personnel will be blinded to treatment assignments, with the exception of designated unblinded team members. Chemoradiotherapy will be administered to all participants and will be open-label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Pembrolizumab + Chemotherapy + Radiotherapy (Experimental): Participants receive pembrolizumab plus one of three chemotherapy regimens chosen by investigator, plus one of three radiotherapy regimens chosen by investigator.
  Interventions: Drug: Pembrolizumab; Radiation: Conventional Radiotherapy (Bladder only); Radiation: Conventional Radiotherapy (Bladder and pelvic nodes); Radiation: Hypofractionated Radiotherapy (Bladder only); Drug: Cisplatin; Drug: Fluorouracil (5-FU); Drug: Mitomycin C (MMC); Drug: Gemcitabine
- Placebo + Chemotherapy + Radiotherapy (Placebo Comparator): Participants receive placebo to pembrolizumab plus one of three chemotherapy regimens chosen by investigator, plus one of three radiotherapy regimens chosen by investigator.
  Interventions: Radiation: Conventional Radiotherapy (Bladder only); Radiation: Conventional Radiotherapy (Bladder and pelvic nodes); Radiation: Hypofractionated Radiotherapy (Bladder only); Drug: Cisplatin; Drug: Fluorouracil (5-FU); Drug: Mitomycin C (MMC); Drug: Gemcitabine; Drug: Placebo to Pembrolizumab

INTERVENTIONS:
Drug: Pembrolizumab — 400 mg of IV (intravenous) pembrolizumab once every 6 weeks.
  Other Names: MK-3475; KEYTRUDA®
  Arms: Pembrolizumab + Chemotherapy + Radiotherapy
Radiation: Conventional Radiotherapy (Bladder only) — 64 Gy of radiation administered to participant's bladder only. Thirty-two fractions will be administered over 6.5 weeks.
Radiation: Conventional Radiotherapy (Bladder and pelvic nodes) — 64 Gy of radiation administered to participant's bladder and pelvic nodes. Thirty-two fractions will be administered over 6.5 weeks.
Radiation: Hypofractionated Radiotherapy (Bladder only) — 55 Gy of radiation administered to participant's bladder only. Twenty fractions will be administered over 4 weeks.
Drug: Cisplatin — 35 mg of cisplatin per cubic meter of body volume, administered once weekly via IV infusion.
Drug: Fluorouracil (5-FU) — 5-FU administered via IV infusion at a dose of 500 mg per cubic meter of body volume on Days 1-5 and 22-26.
Drug: Mitomycin C (MMC) — MMC administered via IV infusion at a dose of 12 mg per cubic meter of body volume on Day 1.
Drug: Gemcitabine — Gemcitabine administered via IV infusion at a dose of 27 mg per cubic meter of body volume twice weekly.
Drug: Placebo to Pembrolizumab — Placebo to intravenous (IV) pembrolizumab administered once every 6 weeks.
  Arms: Placebo + Chemotherapy + Radiotherapy

SUMMARY:
Researchers are looking for new ways to treat muscle-invasive bladder cancer (MIBC). MIBC is a type of cancer that has not spread from the muscles in the bladder to other parts of the body.

MIBC is treated by having surgery to remove the bladder (cystectomy). Not all people choose to have surgery and want to keep their bladder using other treatments.

Chemoradiotherapy (CRT)- is a type of non-surgical treatment for MIBC which combines Chemotherapy (a treatment with medicine to destroy cancer cells or stop them growing) and Radiation therapy (a treatment that uses beams of intense energy [like X-rays] to shrink or get rid of tumors).

Pembrolizumab is an immunotherapy, which is a treatment that helps the immune system fight cancer.

A placebo looks like the study medicine but has no study medicine in it. Using a placebo helps researchers better understand if the study medicine works.

The goal of this study is to learn: 1. If a study medicine pembrolizumab given with Chemoradiotherapy (CRT) can help people live longer without their cancer growing, spreading, or coming back compared to placebo given with CRT. 2.About the safety and how well people tolerate CRT alone or in combination with pembrolizumab.

ELIGIBILITY:
Inclusion Criteria:

* Has a histologically confirmed initial diagnosis of muscle-invasive bladder cancer (MIBC) with predominant urothelial histology
* Has clinically nonmetastatic bladder cancer (N0M0)
* Has planned and is eligible to receive chemoradiotherapy (CRT) and one of the protocol-specified radiosensitizing chemotherapy regimens
* Has Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
* Demonstrates adequate organ function
* Male participants are eligible to participate if they agree to the following during the intervention period and for at least 90 days after the last dose of CRT treatment:

  * Refrain from donating sperm
  * Be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis) and agree to remain abstinent; or must agree to use contraception unless confirmed to be azoospermic
* A female participant is eligible to participate if she is not pregnant or breastfeeding, and at least one of the following conditions applies:

  * Is not a woman of childbearing potential (WOCBP)
  * Is a WOCBP and using a contraceptive method that is highly effective (with a failure rate of <1% per year), with low user dependency or be abstinent from heterosexual intercourse as their preferred and usual lifestyle (abstinent on a long term and persistent basis), during the intervention period and for at least 180 days the time needed to eliminate each study intervention after the last dose of study intervention; and agrees not to donate eggs (ova, oocytes) to others or freeze/store for her own use for the purpose of reproduction during this period. The length of time required to continue contraception for each study intervention is as follows: MK-3475 - 120 days and CRT - 180 days

Exclusion Criteria:

* Has the presence of diffuse carcinoma in situ (CIS) (multiple foci of CIS) throughout the bladder
* Has the presence of urothelial carcinoma (UC) at any site outside of the urinary bladder in the previous 2 years except for Ta stage/T1 stage/CIS of the upper tract if the participant has undergone a complete nephroureterectomy
* Has a known additional malignancy that is progressing or has required active therapy within the past 3 years, except basal cell carcinoma of the skin, squamous cell carcinoma of the skin, superficial bladder cancer or other carcinoma in situ that has undergone potentially curative therapy
* Has the presence of bilateral hydronephrosis
* Has limited bladder function with frequency of small amounts of urine (< 30 mL), urinary incontinence, or requires self-catheterization or a permanent indwelling catheter
* Has received prior pelvic/local radiation therapy for any reason or any antineoplastic treatment for muscle-invasive bladder cancer (MIBC). Treatment for non-muscle invasive bladder cancer (NMIBC) with intravesical instillation therapy that was completed ≥28 days prior to randomization is allowed. Prior systemic treatment of NMIBC is not permitted.
* Received prior therapy with an anti-PD-1 (programmed cell death protein 1), anti-PD-L1 (programmed death-ligand 1), or anti-PD-L2 (programmed cell death 1 ligand 2), or with an agent directed to another stimulatory or coinhibitory T-cell receptor (e.g., CTLA-4 [cytotoxic T-lymphocyte-associated protein 4], OX 40, or CD137 [cluster of differentiation 137])
* Has received a live vaccine within 30 days before the first dose of study medication
* Is currently participating in or has participated in a study of an investigational agent or has used an investigational device within 4 weeks before the first dose of study medication
* Has known severe hypersensitivity (≥Grade 3) to the selected chemotherapy regimen, and/or any of their excipients and excipients of pembrolizumab
* Has a diagnosis of immunodeficiency or is receiving chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 7 days before the first dose of study medication
* Has an active autoimmune disease that has required systemic treatment in the past 2 years (ie, with use of disease modifying agents, corticosteroids or immunosuppressive drugs). Replacement therapy (eg, thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered a form of systemic treatment and is allowed
* Has a history of non-infectious pneumonitis that required steroids or has current pneumonitis
* Has an active infection requiring systemic therapy
* Has a known history of human immunodeficiency virus (HIV) infection
* Has a known history of hepatitis B or known active hepatitis C virus infection
* Has a known history of active tuberculosis (TB; Bacillus tuberculosis)
* Has a known psychiatric or substance abuse disorder that would interfere with the participant's ability to cooperate with the requirements of the study
* Has had an allogenic tissue/solid organ transplant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 520 (Estimated)
Dates: Start 2020-05-19 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2031-11-01 (Estimated)

PRIMARY OUTCOMES:
Bladder Intact Event-Free Survival (BI-EFS) | Up to approximately 76 months
  BI-EFS is defined as the time from randomization to any of the following events: residual/recurrent MIBC post-chemoradiotherapy (CRT), nodal or distant metastases as assessed by computerized tomography (CT) and CT urography (CTU) or magnetic resonance urography (MRU) per blinded independent central review (BICR) and/or biopsy results assessed by central pathology review, radical cystectomy, or death due to any cause. If biopsy is not feasible due to participant safety, the imaging alone will be sufficient. The BI-EFS for all participants will be presented.

SECONDARY OUTCOMES:
Overall Survival (OS) | Up to approximately 95 months
  Time from randomization to death due to any cause.
Metastasis-Free Survival (MFS) | Up to approximately 95 months
  MFS is defined as the time from randomization to the first documented occurrence of nodal or distant metastases as assessed by CT and CTU or MRU per BICR and/or biopsy results assessed by central pathology review If biopsy is not feasible due to participant safety, the imaging alone will be sufficient.
Time to Occurrence of Non-Muscle-Invasive Bladder Cancer (NMIBC) | Up to approximately 95 months
  Time to occurrence of low-grade disease, defined as the time from randomization until the development of NMIBC, will be presented.
Number of Participants Who Experienced an Adverse Event (AE) | Up to approximately 95 months
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who experience an AE will be presented.
Number of Participants Who Discontinued Study Intervention Due to an AE | Up to approximately 1 year
  An AE is any untoward medical occurrence in a participant, temporally associated with the use of study treatment, whether or not considered related to the study treatment. The number of participants who discontinue study treatment due to an AE will be presented.
Change from Baseline in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the European Organization for Research and Treatment of Cancer Quality of Life Questionnaire-Core 30 (EORTC QLQ-C30) | Baseline and up to approximately 24 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. The change from baseline in Global Health Status/Quality of Life (EORTC QLQ-C30 Items 29 and 30) combined score will be presented.
Change from Baseline in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Baseline and up to approximately 24 months
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a better quality of life. The change from baseline in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score will be presented.
Change from Baseline in Urinary, Bowel, and Sexual Domains of the Bladder Cancer Index (BCI) | Baseline and up to approximately 24 months
  The BCI is a validated, condition-specific health questionnaire assessing quality of life among participants with bladder cancer. The BCI contains 36 items which assess 3 domains (urinary, bowel, and sexual) with function and bother subdomains. Scores range from 0 to 100 with higher scores corresponding to better functioning and health-related quality of life. The change from baseline in the combined scores of the urinary, bowel, and sexual domains of the BCI will be presented.
Change from Baseline in the Visual Analog Score (VAS) of the European Quality of Life (EuroQoL)-5 Dimensions, 5-level Questionnaire (EQ-5D-5L) | Baseline and up to approximately 24 months
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 cm vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". The change from baseline in EQ-5D-5L VAS will be presented.
Time to Deterioration (TTD) in the Global Health Status/Quality of Life (Items 29 and 30) Combined Score on the EORTC QLQ-C30 | Up to approximately 24 months
  The EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to the questions "How would you rate your overall health during the past week?" and "How would you rate your overall quality of life during the past week?" are scored on a 7-point scale (1=Very Poor to 7=Excellent). A higher score indicates a better overall outcome. TTD in Global Health Status/Quality of Life is defined as the time from baseline to the first onset of a 10 point or greater decrease from baseline in the Global Health Status/Quality of Life (EORTC QLQ-C30 Items 29 and 30) combined score, with or without subsequent confirmation.
TTD in Physical Functioning (Items 1-5) Combined Score on the EORTC QLQ-C30 | Up to approximately 24 months
  EORTC-QLQ-C30 is a 30-item questionnaire developed to assess the quality of life of cancer patients. Participant responses to 5 questions about their physical functioning are scored on a 4-point scale (1=Not at All to 4=Very Much). A higher score indicates a better quality of life. TTD in Physical Functioning (EORTC QLQ-C30 Items 1-5) combined score is defined as the time from baseline (at randomization) to the first onset of a ≥10-point decrease with confirmation by the subsequent visit of a ≥10-point decrease in physical functioning Items 1 to 5 scale scores.
TTD in Urinary, Bowel, and Sexual Domains of the BCI | Up to approximately 24 months
  The BCI is a validated, condition-specific health questionnaire assessing quality of life among participants with bladder cancer. The BCI contains 36 items which assess 3 domains (urinary, bowel, and sexual) with function and bother subdomains. Scores range from 0 to 100 with higher scores corresponding to better functioning and health-related quality of life. TTD in BCI is defined as a 6, 7, and 7 points or greater worsening from baseline for urinary, bowel, and sexual domains, respectively, with or without subsequent confirmation, under a right-censoring rule.
TTD in the VAS of the EQ-5D-5L | Up to approximately 24 months
  The EQ-5D-5L VAS records the respondent's self-rated health on a 10 cm vertical, visual analogue scale. It is rated by the respondent on a scale 0 to 100, with 0 being "the worst health you can imagine" and 100 being "the best health you can imagine". TTD in EQ-5D-5L VAS is defined as the time from baseline to the first onset of a 7 point or greater decrease from baseline in EQ-5D-5L VAS, with or without subsequent confirmation, under a right-censoring rule.
Time to Cystectomy | Up to approximately 95 months
  Time to cystectomy is defined as time from a participant's randomization to date of cystectomy.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC
Locations (126):
- United States (23):
  - Washington Cancer Institute at MedStar Washington Hospital Center ( Site 0041), Washington D.C., District of Columbia
  - Bay Pines VA Medical Center ( Site 0055), Bay Pines, Florida
  - AdventHealth Orlando-AdventHealth Medical Group Hematology & Oncology at Orlandoc ( Site 0004), Orlando, Florida
  - Norton Cancer Institute ( Site 0044), Louisville, Kentucky
  - Pikeville Medical Center ( Site 0009), Pikeville, Kentucky
  - Baltimore VA Medical Center ( Site 0054), Baltimore, Maryland
  - Washington University ( Site 0003), St Louis, Missouri
  - Summit Medical Group Cancer Center ( Site 6008), Florham Park, New Jersey
  - John Theurer Cancer Center at Hackensack University Medical Center ( Site 0005), Hackensack, New Jersey
  - New York Oncology Hematology P.C ( Site 0024), Albany, New York
  - Roswell Park Cancer Institute ( Site 6009), Buffalo, New York
  - Winthrop University Hospital ( Site 0069), Mineola, New York
  - New York University Perlmutter Cancer Center ( Site 0001), New York, New York
  - Fairview Hospital-Moll Cancer Center ( Site 6013), Cleveland, Ohio
  - Cleveland Clinic Main ( Site 0062), Cleveland, Ohio
  - Cleveland Clinic - Hillcrest Hospital-Hillcrest Hospital Cancer Center ( Site 6012), Mayfield Heights, Ohio
  - MidLantic urology ( Site 0070), Bala-Cynwyd, Pennsylvania
  - Saint Francis Cancer Center ( Site 0026), Greenville, South Carolina
  - Carolina Urologic Research Center ( Site 0002), Myrtle Beach, South Carolina
  - Urology San Antonio Research ( Site 6010), San Antonio, Texas
  - Inova Schar Cancer Institute ( Site 6006), Fairfax, Virginia
  - West Virginia University - Charleston Area Medical Center ( Site 6003), Charleston, West Virginia
  - Froedtert and Medical College of Wisconsin ( Site 0022), Milwaukee, Wisconsin
- Australia (5):
  - Liverpool Hospital ( Site 0220), Liverpool, New South Wales
  - GenesisCare North Shore ( Site 0217), St Leonards, New South Wales
  - Monash Medical Centre ( Site 0216), Clayton, Victoria
  - Austin Health ( Site 0218), Heidelberg, Victoria
  - Sir Charles Gairdner Hospital ( Site 0223), Nedlands, Western Australia
- Chile (5):
  - Oncocentro Valdivia ( Site 7055), Valdivia, Los Ríos Region
  - FALP ( Site 7056), Santiago, Region M. de Santiago
  - Bradfordhill-Clinical Area ( Site 7051), Santiago, Region M. de Santiago
  - ONCOCENTRO APYS-ACEREY ( Site 7054), Viña del Mar, Región de Valparaíso
  - Bradford Hill Norte ( Site 7052), Antofagasta
- Czechia (3):
  - Fakultni nemocnice Olomouc ( Site 0559), Olomouc
  - 2. LF UK a FN Motol ( Site 0555), Prague
  - Nemocnice Na Bulovce ( Site 0556), Prague
- Denmark (2):
  - Herlev og Gentofte Hospital. ( Site 0401), Herlev, Capital Region
  - Odense Universitetshospital ( Site 0403), Odense, Region Syddanmark
- Estonia (2):
  - North Estonia Medical Centre Foundation ( Site 0081), Tallinn, Harju
  - Tartu University Hospital ( Site 0079), Tartu, Tartu
- France (4):
  - Institut Sainte Catherine ( Site 0121), Avignon, Provence-Alpes-Côte d'Azur Region
  - CHU Amiens Picardie Site Sud Amiens ( Site 0123), Amiens, Somme
  - Institut Curie ( Site 0112), Paris
  - A.P.H. Paris. Hopital Bichat Claude Bernard ( Site 0115), Paris
- Guatemala (5):
  - Centro de Investigaciones Clinicas de Latinoamerica S.A. - CELAN ( Site 0146), Guatemala City
  - Oncomedica ( Site 0145), Guatemala City
  - Grupo Medico Angeles ( Site 0143), Guatemala City
  - Medi-K Cayala ( Site 0142), Guatemala City
  - Centro Medico Integral De Cancerología (CEMIC) ( Site 0144), Quetzaltenango
- Hungary (5):
  - BAZ Megyei Korhaz. Klinikai Onkologia es Sugarterapias Centrum ( Site 0092), Miskolc, Borsod-Abauj Zemplen county
  - Petz Aladar Megyei Oktato Korhaz ( Site 0099), Győr, Győr-Moson-Sopron
  - Egeszsegugyi Tudomanyos Tanacs Klinikai Farmakologiai Etikai Bizottsaga ( Site 0095), Budapest
  - Debreceni Egyetem Klinikai Kozpont ( Site 0097), Debrecen
  - Somogy Megyei Kaposi Mor Oktato Korhaz ( Site 0091), Kaposvár
- Israel (6):
  - Soroka Medical Center-Oncology ( Site 7031), Beersheba
  - Rambam Health Care Campus-Oncology Division ( Site 0088), Haifa
  - Hadassah Medical Center. Ein Kerem ( Site 0086), Jerusalem
  - Rabin Medical Center ( Site 7032), Petah Tikva
  - Chaim Sheba Medical Center ( Site 0087), Ramat Gan
  - Sourasky Medical Center ( Site 0089), Tel Aviv
- Italy (8):
  - IRCCS Giovanni Paolo II. Ospedale Oncologico ( Site 0193), Bari, Apulia
  - Fondazione Policlinico Universitario Campus Bio-Medico-Radiation Oncology ( Site 7041), Rome, Lazio
  - Fondazione IRCCS Istituto Nazionale dei Tumori di Milano ( Site 0186), Milan, Lombardy
  - AOU Careggi ( Site 0191), Florence
  - Ospedale Civile di Macerata ( Site 0190), Macerata
  - Ospedale San Raffaele ( Site 0194), Milan
  - Azienda Ospedaliero - Universitaria Policlinico di Modena ( Site 0188), Modena
  - Istituto Nazionale Tumori IRCCS Fondazione Pascale ( Site 0192), Napoli
- Japan (6):
  - Hirosaki University Hospital ( Site 0602), Hirosaki, Aomori
  - University of Tsukuba Hospital ( Site 0605), Tsukuba, Ibaraki
  - Osaka Medical and Pharmaceutical University Hospital ( Site 0604), Takatsuki, Osaka
  - Nagasaki University Hospital ( Site 0600), Nagasaki
  - Institute of Science Tokyo Hospital ( Site 0601), Tokyo
  - Tokyo Metropolitan Komagome Hospital ( Site 0606), Tokyo
- Pauls Stradins Clinical University Hospital ( Site 0073), Riga, Latvia
- Malaysia (4):
  - Hospital Universiti Sains Malaysia ( Site 0237), Kubang Kerian, Kelantan
  - Hospital Pulau Pinang ( Site 0239), George Town, Pulau Pinang
  - Hospital Kuala Lumpur ( Site 0238), Kuala Lumpur
  - University Malaya Medical Centre ( Site 0236), Kuala Lumpur
- Netherlands (2):
  - Netherlands Cancer Institute (NKI) ( Site 0183), Amsterdam, North Holland
  - Erasmus MC ( Site 0182), Rotterdam, South Holland
- Poland (3):
  - Szpital Specjalistyczny im. Ludwika Rydygiera w Krakowie ( Site 0153), Krakow, Lesser Poland Voivodeship
  - Mazowiecki Szpital Wojewódzki w Siedlcach ( Site 0154), Siedlce, Masovian Voivodeship
  - Szpital Wojewodzki im. Mikolaja Kopernika ( Site 0152), Koszalin, West Pomeranian Voivodeship
- Portugal (4):
  - Unidade Local de Saude Loures-Odivelas - Hospital Beatriz Angelo ( Site 0303), Loures, Lisbon District
  - Centro Hospitalar e Universitario de Coimbra ( Site 0306), Coimbra
  - Unidade Local de Saude Lisboa Ocidental - Hospital de São Francisco Xavier ( Site 0302), Lisbon
  - Unidade Local de Saude de Santa Maria - Hospital de Santa Maria ( Site 0305), Lisbon
- Puerto Rico (2):
  - Advance Urology and Laparoscopic Center ( Site 0281), Ponce
  - PAN American Center Oncologic ( Site 0280), San Juan, Rio Piedras
- Romania (7):
  - Institutul Oncologic Prof.Dr. Ion Chiricuta Cluj-Napoca ( Site 0249), Cluj-Napoca, Cluj
  - S.C. Radiotherapy Center Cluj S.R.L ( Site 0252), Cluj-Napoca, Cluj
  - S.C. Centrul de Oncologie Sf. Nectarie SRL ( Site 0248), Craiova, Dolj
  - Policlinica Oncomed SRL ( Site 0254), Timișoara, Timiș County
  - MEMORIAL HEALTHCARE INTERNATIONAL S.R.L. ( Site 0253), Bucharest
  - Institutul Oncologic-Oncologie Medicala ( Site 0256), Cluj-Napoca
  - Institutul Regional de Oncologie Iasi ( Site 0255), Iași
- South Korea (6):
  - National Cancer Center ( Site 0202), Gyeonggi-do, Kyonggi-do
  - Seoul National University Bundang Hospital ( Site 0204), Seongnam-si, Kyonggi-do
  - Asan Medical Center ( Site 0200), Songpagu, Seoul
  - Chungnam National University Hospital ( Site 0203), Daejeon, Taejon-Kwangyokshi
  - Korea University Anam Hospital ( Site 0205), Seoul
  - Severance Hospital Yonsei University Health System ( Site 0201), Seoul
- Spain (3):
  - Instituto Catalan de Oncologia - ICO ( Site 0103), L'Hospitalet de Llobregat, Barcelona
  - Hospital La Fe de Valencia ( Site 0105), Valencia, Valenciana, Comunitat
  - HOSPITAL UNIVERSITARIO VIRGEN DEL ROCIO-Medical Oncology ( Site 0106), Seville
- Turkey (Türkiye) (7):
  - University of Health Sciences,Gulhane School of Medicine-Oncology ( Site 0509), Ankara
  - Ankara Universitesi Tip Fakultesi. ( Site 0502), Ankara
  - Istanbul Uni. Cerrahpasa Tip Fakultesi ( Site 0501), Istanbul
  - T.C. Saglik Bakanligi Turkiye Kamu Hastaneleri Kurumu - Baki-Istanbul Bakirkoy Sadi Konuk Training (, Istanbul
  - Göztepe Prof. Dr. Süleyman Yalçın Şehir Hastanesi-oncology ( Site 0504), Istanbul
  - Ege University Medical Faculty ( Site 0508), Izmir
  - Karadeniz Teknik Universitesi Tip Fakultesi ( Site 0503), Trabzon
- Ukraine (6):
  - Clinical oncology dispensary of Dnipro ( Site 0133), Dnipro, Dnipropetrovsk Oblast
  - Grigoriev Institute for medical Radiology NAMS of Ukraine ( Site 0139), Kharkiv, Kharkivs’ka Oblast’
  - MNPE Regional Center of Oncology ( Site 0134), Kharkiv, Kharkivs’ka Oblast’
  - Ukranian Center of TomoTherapy ( Site 0140), Kropyvnytskiy, Kirovohrad Oblast
  - SNPE National Cancer Institute ( Site 0136), Kyiv, Kyivska Oblast
  - Kyiv City Clinical Oncology Center ( Site 0135), Kyiv
- United Kingdom (7):
  - Betsi Cadwaladr University Health Board ( Site 0447), Rhyl, Denbighshire
  - South Devon Healthcare Foundation Trust. Torbay Hospital ( Site 0444), Torquay, Devon
  - Royal Preston Hospital ( Site 0449), Preston, Lancashire
  - University College London Hospitals NHS Foundation Trust ( Site 0445), London, London, City of
  - The Royal Marsden NHS Foundation Trust. ( Site 0442), London, London, City of
  - Nottingham University Hospital NHS Trust ( Site 0250), Nottingham, Nottinghamshire
  - Darlington Memorial Hospital NHS Trust ( Site 0446), Darlington

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- See also: Merck Clinical Trials Information — https://merckclinicaltrials.com
- See also: Plain Language Summary — https://msd.trialsummaries.com/Study/StudyDetails?id=26156&tenant=MT_MSD_9011